CLINICAL TRIAL: NCT05122000
Title: How Integrity of the Connectome and Nutritional Status Change Brain Function in Breast Cancer Patients Undergoing Chemotherapy
Brief Title: Brain Imaging, Nutrition, and Cognition in Breast Cancer Survivors
Acronym: BRINC
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Tonya Orchard, Associate Professor, Ohio State University
Other Study IDs: 2021C0128
Record Dates: First submitted 2021-11-08; First posted 2021-11-16 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Chemotherapy; Cognitive impairment; Breast cancer survivor; Diet
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood dried blood spots; whole blood venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Up to 78% of women diagnosed with breast cancer experience impairments in their cognitive function (e.g., frequent forgetfulness, slow processing speeds, and difficulties in concentration, multitasking and/or word retrieval) in the course of cancer treatment. These cognitive impairments (CI) have negative effects on patients' social relationships, overall life satisfaction, and treatment adherence. Dietary intake may be an important factor in mitigating risk of CI that breast cancer patients experience. Several studies have suggested that dietary intake of specific nutrients and foods (e.g., carotenoids, B-vitamin, and omega-3 fatty acids rich foods) can be helpful to decrease the severity of cancer-related cognitive impairment (CRCI). High-quality dietary patterns can be also helpful to protect white matter volume and its integrity; damage to and changes in white matter contributes to CRCI. However, despite the high incidence of CRCI in breast cancer patients, very little is known about etiology of CRCI. Thus, the purpose of this observational study with cross-sectional design is to examine the relationships of diet with brain structural and functional outcomes of breast cancer patients. The study will aim to enroll 30 female postmenopausal breast cancer survivors (age 45-75) who have recently completed chemotherapy treatment within 3-12 months from study enrollment. Participants will complete study questionnaires online, and will have an in-person study visit to complete a functional magnetic resonance imagine (MRI) scan, cognitive testing, and blood sample collection via fingerstick and venous blood draw. It is expected that this study will advance the field's understanding and ability to early assess, manage, and prevent CRCI.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III breast cancer diagnosis
* Between 3-12 months post-treatment with anthracycline or taxane-based chemotherapy
* Postmenopausal (at least 12 months without menses; OR on ovarian suppression medication; OR status post oophorectomy)
* English speaking

Exclusion Criteria:

* Women who have permanent ferromagnetic metal in the body, a pacemaker, or have severe claustrophobia
* Women who are pregnant or breastfeeding
* Diagnosis of dementia, psychosis, alcohol or substance use disorders
* Concurrent other malignancy or metastatic malignancy of any kind
* Unable to give informed consent.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer survivors from the Central Ohio area, including those who were seen at The Ohio State University Wexner Medical Center James Cancer Hospital for cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluate feasibility through recruitment and retention | Two years
  Retention is determined by numbers of participants who drop out from the study versus compared to those who complete the study.

SECONDARY OUTCOMES:
Assessment of Brain connectivity | one day
  Assess brain connectivity from MRI images
Assessment of Diet Quality Measures | one day
  Assess diet quality measures from an electronic food frequency questionnaire
Assessment of cognition using the Hopkins Verbal Learning Test | One day
  Assess cognition by using the Hopkins Verbal Learning Test (HVLT), a brief cognitive test of episodic memory and verbal learning.
Assessment of cognition using the WAIS-IV Digit Span | One day
  Assess cognition by using the Wechsler Adult Intelligence Scale (WAIS)-IV Digit Span, a cognitive test of attention and working memory.
Assessment of cognition using the Oral Trail Making Test | One day
  Assess cognition by using the Oral Trail Making Test (TMT), a brief cognitive test of executive function and attention.
Assessment of cognition using the COWA Test | One day
  Assess cognition by using the Controlled Oral Word Association (COWA) Test, a brief cognitive test of oral fluency and executive function.
Assessment of cognition using the Boston Naming Test | One day
  Assess cognition by using the Boston Naming Test Short Form, a brief test of language.
Assessment of presence of CRCI symptoms | One day
  Assess presence of cancer-related cognitive impairment (CRCI) symptoms using the Neuro-QoL Cognitive Function Test, a self-report measurement of cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya S Orchard, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No